CLINICAL TRIAL: NCT01768780
Title: Efficacy of Peripheral Nerve Stimulator in Assessing Sensory Nerve Block Level of Spinal Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4-2012-0692
Record Dates: First submitted 2013-01-08; First posted 2013-01-15 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Orthopedic Surgery-lower Leg Surgery
Keywords: spinal anesthesia; peripheral nerve stimulator; sensory block level

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sensory nerve block level of spinal anesthesia (Experimental): This test group and the control group. Because within the group in two ways to check the level after spinal anesthesia will be.
  Interventions: Device: the anticholinergic glycopyrrolate 0.1 ㎎ + 0-15 mg hyperbaric bupivacaine

INTERVENTIONS:
Device: the anticholinergic glycopyrrolate 0.1 ㎎ + 0-15 mg hyperbaric bupivacaine — The study subjects were patients with planned orthopedic surgery on the infrapatellar area with spinal anesthesia, and 58 patients were recruited sequentially.
  A blood pressure machine, electrocardiogram, and pulse oximeter were connected to the patient in the operating room, and measurements were carried out every 5 minutes. Prior to the induction of anesthesia, the anticholinergic glycopyrrolate 0.1 ㎎ was intravenously administered after the confirmation of intravenous line opening status.
  For spinal anesthesia, the patient was arranged in the lateral recumbent position, and then the L 3-4 area was disinfected. Depending on the surgical region, height, and weight of each patient, 10-15 mg hyperbaric bupivacaine was administered through a 25 G needle.

SUMMARY:
Various methods are used to assess the level of anesthesia block after spinal anesthesia. Among them, ice cubes, alcohol swabs, and needles are commonly used in the clinical setting, but ice is limited by difficulties with management and transportation, and needle assessment has problems owing to the risk of pain, infection, and injury to the patient.

Hence, the alcohol swab is commonly used in practice. However, the absence of pain is more important in the surgical process, and assessing the pain block level is more feasible in practice than assessing the sensory nerve block level using the alcohol swab.

Therefore, it seems to be better to use the peripheral nerve stimulator for the accurate assessment of the pain block level. This has the advantage of continuous measurement of the block level, which can be used in a practical manner in conjunction with the surgical incision.

Hence, the author compared the conventional method using the alcohol swab with the use of the peripheral nerve stimulator to determine which method is more practical in the measurement of spinal anesthesia block level.

ELIGIBILITY:
Inclusion Criteria:

* The study subjects were adult patients, 20-65 years old, who were going to have orthopedic surgery on the infrapatellar area with spinal anesthesia planned and who fell under the American Society of Anesthesiologist physical status classifications of 1 or 2.

Exclusion Criteria:

* Patients who could not read or understand the consent materials or who had pregnancy, hypertension, diabetes, a defect in blood coagulation, cardiovascular disease, or administration of cardiovascular medications were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2012-12; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy of peripheral nerve stimulator as checking sensory block level after spinal anesthesia | Changes of sensory block level at 5 minutes, 10 minutes, 15 minutes, 20 minutes after pinal anesthesia
  The spinal anesthesia block levels were assessed and recorded using the alcohol swab and peripheral nerve stimulation, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea